CLINICAL TRIAL: NCT02110004
Title: Picasso NAV High-Density Mapping Catheter for Signal Analysis of Complex Arrhythmias - First-In-Man
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PIC-152
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ablation procedure (Other): Collect intra-cardiac signals
  Interventions: Procedure: Ablation procedure; Device: Picasso NAV Catheter

INTERVENTIONS:
Procedure: Ablation procedure — The primary purpose of the First-In-Man clinical investigation is to assess the Picasso NAV Catheter's ability to collect intra-cardiac signals within the desired chambers (atrial and/or ventricle) in the heart for the analysis of complex arrhythmias.
Device: Picasso NAV Catheter

SUMMARY:
The primary purpose of the First-In-Man clinical investigation is to assess the Picasso NAV Catheter's ability to collect intracardiac signals within the desired chambers (atrial and/or ventricle) in the heart for the analysis of complex arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation in this clinical investigation.

1. Age > 18 years or older.
2. Patients who have signed the Patient Informed Consent Form (ICF)
3. Patients who are scheduled to undergo a clinically-indicated catheter ablation procedure for the management of a complex arrhythmia. (Patients having undergone a previous ablation procedure may be included.)
4. Subjects who have failed at least one antiarrhythmic drug (AAD) (including AV nodal blocking agents such as beta blockers and calcium channel blockers) as evidenced by recurrent symptomatic complex arrhythmia, or intolerable to the AAD
5. Complex arrhythmias (including atrial fibrillation, atypical flutter, ventricular tachycardia) defined as patients who have been diagnosed with a complex arrhythmia anytime within the last 5 years prior to enrolment. Symptoms may include, but are not restricted to, palpitations, shortness of breath, chest pain, fatigue, left ventricular dysfunction, or other symptoms, or any combination of the above.
6. At least one episode of the complex arrhythmia must have been documented by ECG, Holter, loop recorder, telemetry, implanted device, or transtelephonic monitoring within 12 months of enrollment.
7. Able and willing to comply with all pre-, post-, and follow-up testing and requirements.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not eligible for enrollment.

1. A complex arrhythmia secondary to a reversible cause.
2. Atrial arrhythmias: patients with a left atrial size >55 mm (echocardiography, parasternal long axis view).
3. Left Ventricular Ejection Fraction < 25%
4. NYHA Class III or IV
5. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
6. Atrial arrhythmias: patients with structural atrial disease such as a prior history of atriotomy from prior atrial surgery, presence of an atrial septal defect, and/or presence of an atrial septal closure patch.
7. History of or current blood clotting or bleeding abnormalities, contraindication to systemic anticoagulation (i.e., heparin, warfarin, dabigatran, or a direct thrombin inhibitor)
8. Subjects that have ever undergone valvular cardiac surgical procedure (ie, ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve)
9. Any cardiac surgery within the past 60 days (2 months) (includes PCI)
10. Concurrent enrollment in a study evaluating another device or drug.
11. A complex arrhythmia secondary to electrolyte imbalance, thyroid disease, or non-cardiac cause.
12. Presence of intra-cardiac thrombus or myxoma, interatrial baffle or patch, tumor or other abnormality that precludes catheter introduction or manipulation.
13. Presence of a condition that precludes vascular access.
14. Women of child bearing potential whom are pregnant, lactating, or planning to become pregnant during the course of the clinical investigation
15. Active illness or active systemic infection or sepsis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Intra-procedural investigational device success | Intra-procedure
  Intra-procedural investigational device success
  * Ability to deploy the Picasso NAV Catheter within the atria and/or ventricles
  * The collection of intra-cardiac signals in the atria and/or ventricles
  Measured by number and percentage of physicians able to deploy and collect intra-cardiac signals as outlined in the protocol

SECONDARY OUTCOMES:
Characterize the ideal workflow | Intra-procedure
  Characterize the ideal workflow (defined as catheter preparation, connectivity, and configuration) and the use of the Picasso NAV Catheter's ability to map areas of interest
  Measured by survey questions
Visualize the device | Up to 3 months
  Ability to visualize the device
  Measured by survey questions
Overall safety | Up to 7 days
  Overall safety
  * Primary Adverse Events
  * Procedural complications
  Measured by number and percentage of patients experiencing those adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tom De Potter, Principal Investigator — OLV Hospital; Petr Neuzil, Principal Investigator — Na Homolce Hospital